CLINICAL TRIAL: NCT02236546
Title: FDG-PET/CT as a Biomarker for Treatment Response in Advanced Melanoma
Brief Title: FDG-PET in Advanced Melanoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Yankeelov, Ingram Professor of Cancer Research, Professor of Radiology and Radiological Sciences, Biomedical Engineering, Physics, and Cancer Biology, Director of Cancer Imaging Research, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC MEL 1372; NCI-2014-00179 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC MEL 1372 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
Keywords: fluorodeoxyglucose; FDG; PET/CT; melanoma; imaging biomarkers; cancer imaging
MeSH Terms: conditions — Melanoma | interventions — Immunohistochemistry; Gene Expression; Tissue Array Analysis; Positron-Emission Tomography; Tomography, Emission-Computed; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG-PET/CT (Experimental): Patients undergo [18F]fluorodeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) up to 2 weeks prior to first dose of therapy, after completion of the first treatment course (day 21), and after completion of the fourth treatment course (day 84). Molecular assays on biopsied tissue obtained from a subset of patients will also undergo molecular assays, the results from which will be correlated with FDG-PET/CT data.
  Interventions: Diagnostic Test: [18F]fluorodeoxyglucose; Other: Molecular assays on biopsied tissue; Device: positron emission tomography; Device: computed tomography

INTERVENTIONS:
Diagnostic Test: [18F]fluorodeoxyglucose — FDG is administered intravenously approximately 60 minutes prior to the start of PET image acquisition.
  Other Names: 18-F-deoxy-glucose; 18-F-deoxyglucose; FDG; fluorodeoxyglucose F-18
Other: Molecular assays on biopsied tissue — Correlative studies
  Other Names: immunohistochemistry; genetic assay; laboratory biomarker analysis; molecular profiling; gene expression; tissue microarray
Device: positron emission tomography — Undergo FDG-PET/CT
  Other Names: PET; PET scan; tomography, emission computed
Device: computed tomography — CT that is part of FDG-PET/CT is a low-milliampere, low-resolution scan that is used for anatomic localization and attenuation correction for PET images.
  Other Names: CT; tomography, computed

SUMMARY:
This clinical trial studies how well FDG-PET/CT measures early response in patients with stage III-IV melanoma who are receiving chemotherapy. Positron emission tomography (PET)/computed tomography (CT) uses a metabolic imaging radiotracer, [18F]fluorodeoxyglucose (FDG), which selectively accumulates in tumors. FDG-PET/CT of advanced melanoma before, during, and after treatment may improve methods for predicting which patients may benefit from therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate treatment-induced changes in FDG uptake with changes in tumor size and progression-free survival (PFS) in patients receiving therapy for advanced melanoma.

II. To correlate treatment-induced changes in FDG uptake with changes in the activity and/or expression of available molecular biomarkers from patients receiving therapy for advanced melanoma.

OUTLINE:

Patients undergo FDG-PET/CT up to 2 weeks prior to first dose of therapy, after completion of the first treatment course (day 21), and after completion of the fourth treatment course (day 84).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed Institutional Review Board (IRB)-approved informed consent documentation
* Subjects must be diagnosed with histologically proven stage IV (metastatic) melanoma or stage III with bulky disease which may or may not be amenable for surgery and are receiving therapy at present
* Subjects must be scheduled to begin treatment through the Vanderbilt-Ingram Cancer Center (VICC) Melanoma Program; this will include patients receiving standard-of-care chemotherapy, targeted therapy, and/or immunotherapy, as well as patients accrued to VICC clinical trials for the study of investigational agents
* Subjects must have measurable disease by CT or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria; to comply with PET Response Criteria in Solid Tumors (PERCIST) criteria, subjects should have at least one lesion measuring at least 2 cm in the longest diameter

Exclusion Criteria:

* Subjects who are pregnant or nursing; urine pregnancy test/or serum human chorionic gonadotropin (HCG) will be performed on women of child bearing potential
* Subjects who have experienced allergic or other adverse reactions in response to intravenous injection of fluorinated radiotracers and other contrast media used in PET/CT
* Subjects incapable of giving informed written consent, for the following reasons:

  * Inability to adhere to the experimental protocols for any reason
  * Inability to communicate with the research team
  * Limited ability to give informed consent due to mental disability, altered mental status, confusion, or psychiatric disorders
  * Prisoners or other individuals deemed to be susceptible to coercion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Yankeelov, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to this trial at Vanderbilt Medical Center in Nashville, TN from November 2014 to November 2015
Pre-assignment Details: Four people consented to participate in this trial, one was determined to be ineligible.
Period: Overall Study
Arm/Group | FDG-PET/CT
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FDG-PET/CT
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.66667 (19.85783)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Sum of the Longest Dimension of Target Lesions, Defined by RECIST
Description: The primary imaging metric is percent change in average FDG standardized uptake value (SUV) among the same target lesions between baseline and images acquired after completion of cycle 1. The relationship between tumor SUV change and size change will be assessed using standard linear regression.
Time Frame: Baseline to the completion of 6 courses of treatment
Population: Due to loss of funding data were not collected
Arm/Group | FDG-PET/CT
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response (OR)
Description: The ability of the percent change in average standardized FDG uptake to predict OR will be assessed using the proportional odds model.
Time Frame: Day 84
Population: Due to loss of funding data were not collected
Arm/Group | FDG-PET/CT
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Cox (proportional hazards) regression will be used to assess the association between the percent change in average standardized FDG uptake and PFS.
Time Frame: Time from first treatment until objective tumor progression or death for any reason, assessed up to 7 years
Population: Due to loss of funding data were not collected
Arm/Group | FDG-PET/CT
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Tumor [18F]Fluorodeoxyglucose (FDG) Accumulation
Description: The association between the changes in tumor FDG accumulation with a panel of immunohistochemical biomarkers will be assessed with the Spearman correlation statistic. 95% confidence intervals will be calculated for each variable. Paired changes in biomarker expression between biopsied (i.e., baseline) and biopsy samples will be compared using the nonparametric Wilcoxon signed rank test. Change in binary expression will be compared using McNemar's test. The Wilcoxon rank sum test (or Kruskal Wallis test for more than 2 groups) will be used to compare continuous and ordinal variables.
Time Frame: Baseline to day 21
Population: Due to loss of funding data were not collected
Arm/Group | FDG-PET/CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | FDG-PET/CT
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes